CLINICAL TRIAL: NCT02192307
Title: Effectiveness of Two Water-Based Potassium Oxalate Desensitizers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014047
Record Dates: First submitted 2014-07-14; First posted 2014-07-16 (Estimated); Results first posted 2019-11-05 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-10

CONDITIONS: Dentin Sensitivity
Keywords: Sensitivity
MeSH Terms: conditions — Dentin Sensitivity; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- potassium oxalate gel (Experimental): Professional application
  Interventions: Device: Potassium oxalate
- Potassium oxalate liquid (Active Comparator): Professional application
  Interventions: Device: Potassium oxalate

INTERVENTIONS:
Device: Potassium oxalate
  Other Names: Professional application

SUMMARY:
This study will compare the safety and effectiveness of two water-based potassium oxalate desensitizers on existing dentinal hypersensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent to participate in the study
* Be at least 18 years of age
* Be in good general health, as determined by the Investigator/designee based on review of the health history/update for participation in the study
* Agree to refrain from participating in any other oral/dental product studies for the duration of the study
* Agree to refrain from receiving any elective dentistry (including dental prophylaxis) for the duration of the study
* Agree to refrain from using any oral hygiene products other than the assigned study products for the duration of the study
* Agree to comply with study/product usage instructions; and
* Have at least one tooth with gingival recession and hypersensitivity evidenced by a score of ≥ 1 on the Cold Air Sensitivity Schiff scale during screening

Exclusion Criteria:

* Gross oral neglect or urgent dental treatment needs
* Severe periodontal disease and/or generalized mobility
* Active treatment for periodontitis
* Any disease or condition that could be expected to interfere with examination procedures or safe completion of the study
* Self-reported pregnancy or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts University School of Dental Medicine, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Dipotassium Oxalate Gel: Professional application
  DiPotassium oxalate
- Oxalic Acid Potassium Salt Liquid: Professional application
  Oxalic Acid Potassium Salt Liquid
Period: Overall Study
Arm/Group | Dipotassium Oxalate Gel | Oxalic Acid Potassium Salt Liquid
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Potassium Oxalate Gel: Professional application
  Potassium oxalate gel
- Potassium Oxalate Liquid: Professional application
  Potassium oxalate liquid
- Total: Total of all reporting groups
Arm/Group | Potassium Oxalate Gel | Potassium Oxalate Liquid | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (11.62) | 45.5 (10.82) | 47.5 (11.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 14 | 15 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 1 | 2 | 3
  American Indian | 1 | 0 | 1
  Asian Indian | 2 | 4 | 6
  Asian Oriental | 3 | 1 | 4
  Black | 10 | 12 | 22
  Caucasian | 12 | 10 | 22
  Multiracial | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Air Challenge
Description: The Schiff Sensitivity Scale was assessed for each test tooth via an evaporative air challenge. The examiner recorded the Schiff Index score corresponding to the response to the air challenge. The Schiff Index Sensitivity scale is scored as follows- 0: tooth/subject did not respond to stimulus, 1: tooth/subject responds to stimulus, but does not request discontinuation of stimulus, 2: tooth/subject responds to stimulus and requests discontinuation or moves form stimulus, 3: tooth/subject responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus. The higher the Schiff score, the more sensitive the tooth. The mean change from Baseline was calculated for this measure.
Time Frame: 30 days
Population: Sixty (60) subjects received study products. Sixty (60) subjects completed the study.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Potassium Oxalate Gel; Potassium Oxalate Liquid: Professional application
  Potassium oxalate
Arm/Group | Potassium Oxalate Gel | Potassium Oxalate Liquid
Number analyzed (Participants) | 30 | 30
units on a scale | -0.98 (0.38) | -0.97 (0.47)

2. Secondary Outcome: Change From Baseline Visual Analog Scale
Description: Visual Analog Scale (VAS) - subjects are asked to look at a VAS and designate the level of hypersensitivity they experienced as a result of the thermal and water challenges using a continuum scale of 0 = No tooth pain up to 100 = Worst tooth pain ever experienced.
Time Frame: 30 Days
Population: Sixty (60) subjects received study products. Sixty (60) subjects completed the study.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Potassium Oxalate Gel | Potassium Oxalate Liquid
Number analyzed (Participants) | 30 | 30
units on a scale | -38.10 (27.15) | -32.62 (23.87)

ADVERSE EVENTS:
Time Frame: 30 Days
Arm/Group | Potassium Oxalate Gel | Potassium Oxalate Liquid
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other